CLINICAL TRIAL: NCT03421106
Title: A Multilevel Intervention in the Hunger Relief Network to Improve Diet Among Adults Experiencing Food Insecurity
Acronym: SuperShelf
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection was halted prematurely due to COVID-19.
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Caitlin Caspi, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H20-0076
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-05

CONDITIONS: Food Selection
Keywords: Food insecurity; Food pantries
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Food Pantries (Experimental): Food pantries will transform to offer healthier and more appealing food ; the effect on clients will be measured.
  Interventions: Behavioral: Intervention Food Pantries
- Control Food Pantries (Active Comparator): Food pantries will make no changes during the evaluation period; the effect on clients will be measured.
  Interventions: Other: Control Food Pantries

INTERVENTIONS:
Behavioral: Intervention Food Pantries — Food pantries will receive consulting services to transform their food offerings and environment in order to influence client health behaviors.
  Arms: Intervention Food Pantries
Other: Control Food Pantries — Normal food pantry use
  Arms: Control Food Pantries

SUMMARY:
The investigator proposes an evaluation of a randomized, sustainable intervention in 8 intervention and 8 control pantries. We will enroll a sample clients at the food pantry at baseline and follow them for 1 year to assess changes in overall diet quality (the primary outcome) and cardiovascular health. We will also enroll a sample of clients at follow-up to assess to assess the nutritional quality of food selected at the pantry.

DETAILED DESCRIPTION:
Evaluate the health impact of an intervention targeting the hunger relief network and the clients with food insecurity it serves. The long-term goal of this work is to reduce nutrition-related health disparities by intervening on a system that serves individuals at high risk for chronic disease. In 2014, an estimated 14% of U.S. households experienced food insecurity (i.e., they lacked access to enough food for an active, healthy life for all household members). Large numbers of low-income, racial/ethnic minority, and immigrant families who experience food insecurity rely on a hunger relief network that includes food banks and food pantries. Pantry clients have demonstrated poor nutritional outcomes, high chronic disease rates, and dissatisfaction with the quality and cultural-appropriateness of food offered. Unlike other food assistance programs, there are currently no standards on the nutritional quality of pantry offerings, but recent work by our study team demonstrated the need to improve the healthfulness of hunger relief network inventory. We proposed an evaluation of a randomized, sustainable intervention in 8 intervention and 8 control pantries. We will enroll clients at baseline and follow them for 1 year to assess changes in overall diet quality (the primary outcome). Working with our food bank partners, the intervention at the pantry level targets the supply of nutritious foods. At the client level, the intervention targets healthy food demand. Measured outcomes include overall diet quality (the primary outcome), as assessed by the Healthy Eating Index-2015 (HEI), the nutritional quality of foods selected at the food shelf visit, and cardiovascular disease health (assessed by the American Heart Association's Life's Simple 7 scores). The study will also evaluate the impact of a multilevel intervention on the nutritional quality of pantry offerings. The study also aims to improve implementation of practices that promote a nutrition-focused hunger relief network.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years old

* Mentally capable of consent and participation
* Speak English, Spanish, or Somali
* Have access to a phone

Exclusion Criteria:

* Not capable of consent or participation
* Speak only languages other than English, Spanish or Somali
* Not a food pantry user

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin E Caspi, ScD, Principal Investigator — University of Connecticut
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Caspi C, Gordon N, Bliss Barsness C, Bohen L, Canterbury M, Peterson H, Wolfson J, Pratt R. A randomized study of food pantry environment-level change following the SuperShelf intervention. Transl Behav Med. 2022 Jul 7;12(6):764-774. doi: 10.1093/tbm/ibac003. PMID 35666208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two samples of participants were enrolled. The first (Sample A, n=317), had measures collected at two time points. They were enrolled at baseline and followed for one year to assess change in diet quality (primary outcome) and cardiovascular measures (secondary outcome). The second (Sample B, n=187) had measures collected at one time point only. They were enrolled at the pantry during the follow-up period to assess post-intervention client cart diet quality (secondary outcome).
Groups:
- Intervention Food Pantries and Clients: Food pantries will transform to offer healthier and more appealing food; the effect on clients will be measured;
  Intervention Food Pantries: Food pantries will receive consulting services to transform their food offerings and environment in order to influence client health behaviors.
  Intervention Clients: Clients who use and were recruited at intervention food pantries.
- Control Food Pantries and Clients: Food pantries will make no changes during the evaluation period; the effect on clients will be measured.
  Control Food Pantries: Normal food pantry operations during the evaluation period.
  Control Clients: Clients who use and were recruited at control food pantries.
Period: Sample A (Followed for 1 Year)
Arm/Group | Intervention Food Pantries and Clients | Control Food Pantries and Clients
Started | 158 | 159
Completed | 102 | 105
Not Completed | 56 | 54
Period: Sample B (Evaluated at Post Only)
Arm/Group | Intervention Food Pantries and Clients | Control Food Pantries and Clients
Started | 85 | 102
Completed | 85 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Food Pantries and Clients: Food pantries will transform to offer healthier and more appealing food; the effect on clients will be measured;
  Intervention Food Pantries: Food pantries will receive consulting services to transform their food offerings and environment in order to influence client health behaviors;
  Intervention Clients: Clients who use and were recruited at intervention food pantries.
- Control Food Pantries and Clients: Food pantries will make no changes during the evaluation period; the effect on clients will be measured;
  Control Food Pantries: Normal food pantry operations during the evaluation period;
  Control Clients: Clients who use and were recruited at control food pantries.
- Total: Total of all reporting groups
Arm/Group | Intervention Food Pantries and Clients | Control Food Pantries and Clients | Total
Number analyzed (Participants) | 243 | 261 | 504
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0
  18-64 | 210 | 227 | 437
  65 years and older | 31 | 31 | 62
  Unknown | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 total participants did not provide binary sex designations.
  Participants
    number analyzed (Participants) | 240 | 258 | 498
    Female | 146 | 169 | 315
    Male | 94 | 89 | 183
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 15 | 35
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 23 | 56 | 79
  White | 146 | 153 | 299
  More than one race | 34 | 19 | 53
  Unknown or Not Reported | 19 | 16 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 243 | 261 | 504

OUTCOME MEASURES:

1. Primary Outcome: Overall Diet Quality of Clients
Description: Assessed by Healthy Eating Index-2015 scores (scale 0-100), with 100 representing the best possible score (i.e., nutritional quality best aligned with Dietary Guidelines for Americans)
Time Frame: Baseline, 1 year
Population: COVID-19 disrupted intervention and post-evaluation activities in 5 sites. The analysis includes participants in Sample A at the 11 completed sites.
Measure: Least Squares Mean (Standard Error); unit: Pre-post change in HEI score on a scale
Arm/Group | Intervention Food Pantries and Clients | Control Food Pantries and Clients
Number analyzed (Participants) | 89 | 104
Pre-post change in HEI score on a scale | 1.09 (1.45) | -1.42 (1.52)
Statistical Analysis 1: Comparison: Intervention Food Pantries and Clients vs Control Food Pantries and Clients; Test type: Superiority; p = 0.23, Mixed Models Analysis; Mean Difference (Net) = 2.53

2. Secondary Outcome: Nutritional Quality of Food Selected by Clients at the Food Pantry
Description: as for outcome 1
Time Frame: 1 year post-sample comparison
Population: COVID-19 disrupted intervention and post-evaluation activities in 5 sites. The analysis includes participants in Sample B at the 11 completed sites.
Measure: Mean (Standard Deviation); unit: Post-sample HEI score
Arm/Group | Intervention Food Pantries and Clients | Control Food Pantries and Clients
Number analyzed (Participants) | 85 | 102
Post-sample HEI score | 60.6 (11.8) | 64.0 (10)

3. Secondary Outcome: Cardiovascular Health
Description: American Heart Association's Life's Simple 7 (LS7) scores (scale 0 -7), with 7 representing the best possible score for cardiovascular health
Time Frame: Baseline, 1 year
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Pre-post change in LS7 score on a scale
Arm/Group | Intervention Food Pantries and Clients | Control Food Pantries and Clients
Number analyzed (Participants) | 89 | 104
Pre-post change in LS7 score on a scale | -0.09 (0.15) | 0.41 (0.16)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the period of follow-up for each participant. In Sample A, the mean follow-up was 13.9 months. In Sample B, there was no follow-up and no monitoring of adverse events.
Arm/Group | Intervention Food Pantries and Clients | Control Food Pantries and Clients
All-Cause Mortality (participants affected / at risk) | 1/158 | 1/159
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/159
Other Adverse Events (participants affected / at risk) | 0/158 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03421106/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT03421106/ICF_001.pdf